CLINICAL TRIAL: NCT06516029
Title: Real-World Evaluation of Patient Characteristics and Treatment Patterns Among Patients With CML-CP Treated With Asciminib (ABL-2022-02)
Brief Title: Real-World Evaluation of Patient Characteristics and Treatment Patterns Among Patients With CML-CP Treated With Asciminib
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CABL001A0US03
Record Dates: First submitted 2024-07-07; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Overall Asciminib Cohort: Adult patients diagnosed with Ph+ CML-CP, with or without the T3151 mutation, who initiated asciminib in any line of therapy.

SUMMARY:
A retrospective, non-interventional cohort study design using data obtained from the Flatiron Health oncology electronic health record (EHR)-derived de-identified database, was used to address the study objectives.

The overall asciminib cohort included adult patients with Philadelphia positive (Ph+) chronic myeloid leukemia (CML) in chronic phase (CML-CP), with or without the T3151 mutation, who initiated asciminib in any line of therapy. The third-line or later (3L+) asciminib cohort included adult patients with Ph+ CML-CP who did not have T315I mutation and initiated asciminib after prior use of at least 2 different tyrosine kinase inhibitors (TKIs) or omacetaxine. The 3L asciminib cohort included the subgroup of the 3L+ asciminib cohort who initiated asciminib after prior use of 2 different TKIs or omacetaxine. The fourth-line or later (4L+) asciminib cohort included the subgroup of the 3L+ asciminib cohort who initiated asciminib after prior use of at least 3 different TKIs or omacetaxine.

ELIGIBILITY:
Inclusion criteria:

* Patients who initiated asciminib as identified by Flatiron through the Flatiron Health-Novartis Scemblix CML Spotlight database study.
* Patients had at least one diagnosis for CML (International Classification of Diseases, 9th Edition, Clinical Modification [ICD-9-CM]: 205.1x; International Classification of Diseases, 10th Edition, Clinical Modification [ICD-10-CM]: C92.1x).
* Diagnosed with CP as identified by Flatiron through chart abstraction.
* Had 2 or more documented clinical visits, on different days in the Flatiron data on or after 1 January 2011.
* Had evidence of treatment with asciminib on or after Food and Drug Administration (FDA) approval date (29 October 2021), with data granularity availability at least at the month level for dates of asciminib use.
* Had CML initial diagnosis date on or after 1 January 2011.
* Had 1 or more clinical activity within 6 months prior to asciminib initiation (e.g., medical visit, medication order, lab test, etc.).

Exclusion criteria:

* Patients who did not meet inclusion criteria listed above.
* Had stem-cell transplant (SCT) on or prior to asciminib initiation or unknown SCT date.
* Diagnosed with CML in accelerated phase (AP) or blast crisis (BC) before asciminib initiation, as identified by Flatiron through chart abstraction, or had blast greater than 15% or unknown blast result within 60 days prior to asciminib initiation.
* Patients had received a clinical study drug between 15 November 2017 and 4 December 2019 (randomization dates for the ASCEMBL trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Age at Index Date | Up to 137 months
  Index date was defined as the date of initiation for asciminib.
Gender at Index Date | Up to 137 months
  Index date was defined as the date of initiation for asciminib.
Race at Index Date | Up to 137 months
  Index date was defined as the date of initiation for asciminib.
Type of Practice at Index Date | Up to 137 months
  Types of practices included: community and academic practices. Index date was defined as the date of initiation for asciminib.
Eastern Cooperative Oncology Group Performance Score (ECOG-PS) at Index Date | Up to 137 months
  ECOG-PS describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores ranged from a lower value of 0 (fully active, able to carry on all pre-disease performance without restriction) up to 4 (completely disabled; cannot carry on any selfcare; totally confined to bed or chair).
  Index date was defined as the date of initiation for asciminib.
Number of Patients Categorized by the Five Most Common Baseline Comorbidities | Baseline
  Baseline was defined as the time between the date of initial CML diagnosis up to (and excluding) the date of asciminib initiation (index date).
Number of Patients Categorized by Last Molecular Response (MR) Achieved Within 3-months Prior to Index Date | Up to 3 months pre-index date
  MR categories included:
  * MR0 (BCR::ABL1 greater than 10%)
  * MR1 (BCR::ABL1 less than or equal to 10%)
  * MR2 (BCR::ABL1 less than or equal to 1%)
  * MR3/Major MR (BCR::ABL1 less than or equal to 0.1%)
  * MR4 or better (BCR::ABL1 less than or equal to 0.01%)
  Index date was defined as the date of initiation for asciminib.
Median Duration of Observation from Index Date to the end of the Study Period | Up to 13 months
  The study period was defined as the time between the index date (inclusive) until the earliest of stem-cell transplant (SCT), death, loss-to-follow-up (i.e., last activity in the electronic medical record data), or end of data availability (i.e., 30 November 2022). The index date was the date of initiation for asciminib.
Number of Patients by First Observed Line of Therapy with Asciminib at Index Date | Up to 137 months
  Index date was defined as the date of initiation for asciminib.
Number of Patients Categorized by Dosage of Asciminib at Index Date | Up to 137 months
  Index date was defined as the date of initiation for asciminib.
Number of Patients by Status at End of First Observed Line of Therapy with Asciminib | From date of asciminib initiation to end of study period, up to 13 months
  Status:
  * Continued asciminib treatment (included dose change/held).
  * Discontinued asciminib treatment.
Number of Patients by Type of First Tyrosine Kinase Inhibitor (TKI) Received Before Asciminib Initiation | Up to 137 months
Number of Patients by Type of TKI Received Immediately Before Asciminib Initiation | Up to 137 months
Number of Patients by Type of TKI Received Anytime Before Asciminib Initiation | Up to 137 months
Number of Patients by Most Common Treatment Sequence | From initial CML diagnosis until the end of study period, up to 143 months
Asciminib Treatment Persistence Rate Post-Index Date | Week 12, week 24 post-index date
  Index date was defined as the date of initiation for asciminib.

SECONDARY OUTCOMES:
Number of Patients Categorized by Best Molecular Response (MR) Achieved Within 12-months Post-index Date | 12 months post-index date
  MR categories included:
  * MR0 (BCR::ABL1 greater than 10%)
  * MR1 (BCR::ABL1 less than or equal to 10%)
  * MR2 (BCR::ABL1 less than or equal to 1%)
  * MR3/Major MR (BCR::ABL1 less than or equal to 0.1%)
  * MR4 or better (BCR::ABL1 less than or equal to 0.01%)
  Index date was defined as the date of initiation for asciminib.
Number of Patients With one or More MR Test Post-index Date who Achieved or Maintained MR3/Major MR (MMR) | Week 12, week 24 post-index date
  MR3/MMR was defined as BCR::ABL1 less than or equal to 0.1%. Index date was defined as the date of initiation for asciminib.
Number of Patients With one or More MR Test Post-index Date who Achieved or Maintained MR2 | Week 12, week 24 post-index date
  MR2 was defined as BCR::ABL1 less than or equal to 1%. Index date was defined as the date of initiation for asciminib.
Number of Patients Without MR3/MMR Prior to Asciminib Initiation who Achieved MR3/MMR Post-index Date | Week 12, week 24 post-index date
  MR3/MMR was defined as BCR::ABL1 less than or equal to 0.1%. Index date was defined as the date of initiation for asciminib.
Median Time to MR3/MMR Post-index Date Among Patients Without MR3/MMR Prior to Asciminib Initiation | From index date until the end of study period, up to 13 months
  MR3/MMR was defined as BCR::ABL1 less than or equal to 0.1%. Index date was defined as the date of initiation for asciminib.
Number of Patients Without MR2 Prior to Asciminib Initiation who Achieved MR2 Post-index Date | Week 12, week 24 post-index date
  MR2 was defined as BCR::ABL1 less than or equal to 1%. Index date was defined as the date of initiation for asciminib.
Median Time to MR2 Post-index Date Among Patients Without MR2 Prior to Asciminib Initiation | From index date until the end of study period, up to 13 months
  MR3/MMR was defined as BCR::ABL1 less than or equal to 1%. Index date was defined as the date of initiation for asciminib.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States